CLINICAL TRIAL: NCT02968368
Title: A Phase 3, Randomized, Placebo Controlled, Prospective, Multicenter Study With Oral Ferric Maltol for the Treatment of Iron Deficiency Anemia in Subjects With Chronic Kidney Disease
Brief Title: Study With Oral Ferric Maltol for the Treatment of Iron Deficiency Anemia in Subjects With Chronic Kidney Disease
Acronym: AEGIS-CKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shield Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST10-01-303
Record Dates: First submitted 2016-08-30; First posted 2016-11-18 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Renal Insufficiency, Chronic; Iron-Deficiency Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency | interventions — ferric maltol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral ferric maltol (Experimental): 30mg capsules BID
  Interventions: Drug: Ferric maltol
- Oral placebo (Placebo Comparator): Matching placebo capsules BID
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ferric maltol
  Other Names: Feraccru
  Arms: Oral ferric maltol
Other: Placebo
  Arms: Oral placebo

SUMMARY:
To evaluate the efficacy of oral ferric maltol compared with placebo in the treatment of IDA in subjects with CKD

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the information given in the Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved information sheet and consent form. Must sign and date the informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations prior to any study mandated procedure.
2. Willing and able to comply with study requirements.
3. Age ≥ 18 years at the time of informed consent.
4. A current diagnosis of CKD with an estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73m2 and ≥15 mL/min/1.73m2, as calculated using the abbreviated version of the Modified Diet in Renal Disease equation (MDRD) assessed via screening laboratory results.
5. Iron deficiency anemia defined by the following criteria assessed via screening laboratory results:

   1. Hb <11.0g/dL and ≥8.0g/dL
   2. AND ferritin <250ng/mL with a Transferrin saturation (TSAT) <25% OR ferritin <500ng/mL with a TSAT of <15%
6. Female subjects of childbearing potential (including perimenopausal females who have had a menstrual period within 1 year prior to screening) must agree to use a reliable method of contraception until study completion and for at least 4 weeks following their final study visit. Reliable contraception is defined as a method which results in a low failure rate, i.e., less than 1% per year when used consistently and correctly, such as implants, injectables, some intrauterine contraceptive devices (IUDs), complete sexual abstinence, a vasectomized partner and oral contraceptive medications. Female subjects who are surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) or postmenopausal (defined as no menstrual period within 1 year of screening) are also allowed to participate.

Exclusion Criteria:

1. Anemia due to any cause other than iron deficiency, including, but not limited to:

   1. Untreated or untreatable severe malabsorption syndrome.
   2. Myelosuppression use (permitted if taken at a stable dose and frequency for at least 12 weeks prior to randomization and are expected to stay stable throughout the double-blind treatment period so long as there is no clinical evidence of the myelosuppression contributing to the subject's anemia).
2. Administration with any of the following prior to randomization:

   1. IV iron injection within the previous 4 weeks or administration of intramuscular or depot iron preparation within the previous 12 weeks.
   2. Single agent oral iron supplementation, taken specifically to treat anemia (e.g. ferrous sulfate, fumarate and gluconate) within the previous 2 weeks. Multivitamins are permitted.
   3. Use if ferric citrate and sucroferric oxyhydroxide within the previous 1 week.
   4. ESAs within the previous 4 weeks
   5. Blood transfusion or donation within the previous 12 weeks.
   6. Dimercaprol or cloramphenicol within the previous 7 days.
   7. Current use of methyldopa.
3. Currently receiving dialysis or initiation of dialysis is considered likely during the study.
4. Renal transplant within 12 months prior to randomization or is considered likely during the study.
5. Known hypersensitivity or allergy to the active substance or excipients of ferric maltol or placebo capsules.
6. Contraindication for treatment with iron preparations, e.g. hemochromatosis, chronic hemolytic disease, sideroblastic anemia, thalassemia, or lead intoxication induced anemia.
7. Impaired liver function as indicated by alanine aminotransferase (ALT) or aspartate transaminase (AST) > 3 times the upper limit of normal as assessed via screening laboratory results.
8. Clinically significant vitamin B12 or folic acid deficiency as determined by the screening laboratory results (retest following at least 2 weeks of starting treatment with vitamin B12 or folate replacement is permitted).
9. Pregnant or breast feeding.
10. Concomitant medical conditions with significant active bleeding likely to initiate or prolong anemia; for example coagulation disorders or recurrent GI bleeding.
11. Scheduled or expected major surgery during the course of the study. (Minor surgeries not associated with significant blood loss, in the Investigator's judgement, are permitted e.g. surgery related to fistulae or vascular access, minor dental extractions, incision and drainage of abscess or simple excisions).
12. Participation in any other interventional clinical study within 30 days prior to screening.
13. Cardiovascular, liver, renal, hematologic, psychiatric, neurologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease that, in the opinion of the Investigator, may adversely affect the safety of the subject and/or efficacy of the study drug or severely limit the lifespan of the subject.
14. Any other unspecified reason that, in the opinion of the Investigator or the Sponsor make the subject unsuitable for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sampson, MBChB, Study Director — Shield Therapeutics
Locations (27):
- United States (27):
  - Peoria, Arizona
  - Phoenix, Arizona
  - Prescott, Arizona
  - Tucson, Arizona
  - La Mesa, California
  - Long Beach, California
  - Roseville, California
  - Sacramento, California
  - Denver, Colorado
  - Coral Springs, Florida
  - Edgewater, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Macon, Georgia
  - Shreveport, Louisiana
  - Pontiac, Michigan
  - Roseville, Michigan
  - Las Vegas, Nevada
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Wilmington, North Carolina
  - Bethlehem, Pennsylvania
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - El Paso, Texas
  - San Antonio, Texas
  - Hampton, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pergola PE, Kopyt NP. Oral Ferric Maltol for the Treatment of Iron-Deficiency Anemia in Patients With CKD: A Randomized Trial and Open-Label Extension. Am J Kidney Dis. 2021 Dec;78(6):846-856.e1. doi: 10.1053/j.ajkd.2021.03.020. Epub 2021 May 23. PMID 34029682

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Ferric Maltol: 30mg capsules BID
  Ferric maltol
- Oral Placebo: Matching placebo capsules BID
  Placebo
Period: Double Blind Phase
Arm/Group | Oral Ferric Maltol | Oral Placebo
Started | 111 | 56
Completed | 90 | 39
Not Completed | 21 | 17
Period: Open Label Phase
Arm/Group | Oral Ferric Maltol | Oral Placebo
Started | 86 | 39
Completed | 67 | 25
Not Completed | 19 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Ferric Maltol | Oral Placebo | Total
Number analyzed (Participants) | 111 | 56 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 19 | 53
  >=65 years | 77 | 37 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (12.43) | 65.2 (12.79) | 67.4 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 39 | 117
  Male | 33 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 14 | 40
  Not Hispanic or Latino | 84 | 42 | 126
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 12 | 35
  White | 81 | 42 | 123
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 111 | 56 | 167

OUTCOME MEASURES:

1. Primary Outcome: Change in Hb Concentration From Baseline to Week 16
Description: Change in hemoglobin concentration from baseline to Week 16.
Time Frame: 16 weeks
Population: ITT
Measure: Least Squares Mean (Standard Deviation); unit: g/dl
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 88 | 40
g/dl | 0.50 (0.122) | -0.02 (0.165)
Statistical Analysis 1: Comparison: Oral Ferric Maltol vs Oral Placebo; Test type: Superiority; p = 0.0149, ANCOVA; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.102 to 0.930], Standard Error of Mean 0.210

2. Secondary Outcome: Number of Subjects That Achieve an Increase in Hb Concentration of ≥1 g/dL at Week 16
Description: Number of subjects that achieve an increase in Hemoglobin concentration of ≥1 g/dL at Week 16
Time Frame: 16 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 111 | 56
Participants | 22 | 5

3. Secondary Outcome: Number of Subjects That Achieve a Hb Concentration of ≥11 g/dL at Week 16
Description: Number of subjects that achieve a Hemoglobin concentration of ≥11 g/dL at week 16
Time Frame: 16 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 111 | 56
Participants | 30 | 7

4. Secondary Outcome: Change in Hb Concentration From Baseline to Week 8
Description: Change in Hemoglobin concentration from baseline to Week 8
Time Frame: 8 weeks
Population: Where a subject had dropped from the study, we used a LOCF by MI methodology to impute values. Therefore the number of subjects and observations at a given time-point may differ.
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 98 | 47
g/dl | 0.53 (0.901) | 0.00 (0.909)

5. Secondary Outcome: Number of Subjects That Achieve an Increase in Hb Concentration of ≥2 g/dL at Week 16
Description: Number of subjects that achieve an increase in Hemoglobin concentration of ≥2 g/dL at Week 16
Time Frame: 16 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 111 | 56
Participants | 7 | 0

6. Secondary Outcome: Changes in Ferritin From Baseline to Week 16
Description: Changes in iron parameter - ferritin - from baseline to week 16
Time Frame: baseline to week 16
Population: ITT OC
Measure: Least Squares Mean (Standard Deviation); unit: ug/l
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 111 | 56
ug/l | 33.13 (6.166) | -5.90 (9.137)
Statistical Analysis 1: Comparison: Oral Ferric Maltol vs Oral Placebo; Test type: Superiority; p = 0.0006, ANCOVA; Mean Difference (Final Values) = 39.03, 95% CI 2-sided [17.070 to 60.992], Standard Error of Mean 11.097

7. Secondary Outcome: Number of Participants With (TEAEs)
Description: Number of Participants with Treatment-Emergent Adverse Events (TEAEs)
Time Frame: Week 16
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 111 | 56
Participants | 75 | 42

8. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs)
Description: Number of Participants with Treatment-Emergent Serious Adverse Events (TESAEs) during the double blind phase
Time Frame: Week 16
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 111 | 56
Participants | 23 | 12

9. Secondary Outcome: Changes in TSAT From Baseline to Week 16
Description: Changes in iron parameters - TSAT - from baseline to week 16
Time Frame: baseline to week 16
Population: ITT OC
Measure: Least Squares Mean (Standard Deviation); unit: TSAT (%)
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 111 | 56
TSAT (%) | 4.32 (0.719) | -0.15 (1.060)
Statistical Analysis 1: Comparison: Oral Ferric Maltol vs Oral Placebo; Test type: Superiority; p = 0.0007, ANCOVA; Mean Difference (Final Values) = 4.46, 95% CI 2-sided [1.928 to 7.001], Standard Error of Mean 1.282

10. Secondary Outcome: Changes in Iron Parameter From Baseline to Week 16
Description: Changes in iron parameters - serum iron - from baseline to week 16
Time Frame: from baseline to week 16
Population: ITT OC
Measure: Least Squares Mean (Standard Deviation); unit: umol/l
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 111 | 56
umol/l | 1.87 (0.397) | 0.01 (0.586)
Statistical Analysis 1: Comparison: Oral Ferric Maltol vs Oral Placebo; Test type: Superiority; p = 0.0098, ANCOVA; Mean Difference (Final Values) = 1.86, 95% CI 2-sided [0.457 to 3.261], Standard Error of Mean 0.708

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) during the open label phase
Time Frame: Week 52
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 86 | 39
Participants | 76 | 35

12. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs)
Description: Number of Participants with Treatment-Emergent Serious Adverse Events (TESAEs) during the open label phase
Time Frame: Week 52
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ferric Maltol | Oral Placebo
Number analyzed (Participants) | 86 | 39
Participants | 27 | 9

ADVERSE EVENTS:
Time Frame: 16 week double blind phase
Description: 167 subjects. Definitions of AEs and SAEs in line with clintrials.gov definitions
Groups:
- Oral Ferric Maltol DB: 30mg capsules BID
  Ferric maltol
  double blind phase
- Oral Placebo DB: Matching placebo capsules BID
  Placebo
  double blind phase
- Oral Ferric Maltol OL: 30mg capsules BID
  Ferric maltol
  open label phase
- Oral Placebo OL: Matching placebo capsules BID
  Placebo
  open label phase
Arm/Group | Oral Ferric Maltol DB | Oral Placebo DB | Oral Ferric Maltol OL | Oral Placebo OL
All-Cause Mortality (participants affected / at risk) | 75/111 | 42/56 | 76/86 | 35/39
Serious Adverse Events (participants affected / at risk) | 23/111 | 12/56 | 27/86 | 9/39
Other Adverse Events (participants affected / at risk) | 75/111 | 42/56 | 76/86 | 35/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Ferric Maltol DB (N=111) | Oral Placebo DB (N=56) | Oral Ferric Maltol OL (N=86) | Oral Placebo OL (N=39)
Sudden death (General disorders) | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Hemorrhagic anemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Duodenal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1 | 2
Hypertensive emergency (Vascular disorders) | 1 | 1 | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Normochromic normocytic anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Necrotizing fasciitis (Infections and infestations) | 0 | 0 | 1 | 0
Streptococcal bacteremia (Infections and infestations) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hemoglobin decreased (Investigations) | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lacunar stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Hypovolemic shock (Vascular disorders) | 0 | 0 | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Ferric Maltol DB (N=111) | Oral Placebo DB (N=56) | Oral Ferric Maltol OL (N=86) | Oral Placebo OL (N=39)
Diarrhea (Gastrointestinal disorders) | 10 | 5 | 7 | 5
Nausea (Gastrointestinal disorders) | 9 | 5 | 10 | 5
Constipation (Gastrointestinal disorders) | 9 | 2 | 14 | 5
Feces discolored (Gastrointestinal disorders) | 8 | 1 | 7 | 1
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 21 | 13 | 25 | 13 — TEAEs in <5% of Subjects Overall by SOC
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 7 | 5 | 6
Infections and infestations (Infections and infestations) | 17 | 13 | 39 | 19 — TEAEs in <5% of Subjects Overall by SOC
Urinary tract infection (Infections and infestations) | 7 | 5 | 7 | 4
Renal and urinary disorders (Renal and urinary disorders) | 10 | 6 | 0 | 0 — TEAEs in <5% of Subjects Overall by SOC
Acute kidney injury (Renal and urinary disorders) | 5 | 4 | 0 | 0
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5 | 9 | 0 | 0 — TEAEs in <5% of Subjects Overall by SOC
Anemia (Blood and lymphatic system disorders) | 4 | 6 | 0 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 45 | 17 | 48 | 18
Vomiting (Gastrointestinal disorders) | 0 | 0 | 7 | 0
General disorders and administration site conditions (General disorders) | 0 | 0 | 16 | 5
Fatigue (General disorders) | 0 | 0 | 6 | 1
Edema peripheral (General disorders) | 0 | 0 | 7 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 5 | 4
Nasopharyngitis (Infections and infestations) | 0 | 0 | 9 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 7 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 8 | 4
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 0 | 0 | 17 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 7 | 1
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 19 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 2
Vascular disorders (Vascular disorders) | 0 | 0 | 16 | 5
Hypertension (Vascular disorders) | 0 | 0 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT02968368/Prot_SAP_000.pdf